CLINICAL TRIAL: NCT03218709
Title: Effect of Multi-vitamins With Minerals on Uric Acid Metabolism in Subjects With Hyperuricemia: A Randomized, Double-blinded, Placebo-controlled Trail
Brief Title: The Intervention of Multi-vitamin With Minerals to Hyperuricemia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Di Li, PhD, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZXYZM-6
Record Dates: First submitted 2017-03-22; First posted 2017-07-14 (Actual); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Hyperuricemia
MeSH Terms: conditions — Hyperuricemia | interventions — Minerals

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High-dose multi-vitamins with minerals (Experimental): Generic name: High-dose multi-vitamins with minerals tablets Dosage form: Capsule Frequency: Two pills daily for 6 months
  Interventions: Combination Product: High-dose multi-vitamins with minerals
- Low-dose multi-vitamins with minerals (Experimental): Generic name: Low-dose multi-vitamins with minerals tablets Dosage form: Capsule Frequency: Two pills daily for 6 months
  Interventions: Combination Product: Low-dose multi-vitamins with minerals
- Hypouricemic tablets (Active Comparator): Generic name: Hypouricemic tablets Dosage form: Capsule Frequency: Six pills daily for 3 months
  Interventions: Combination Product: Hypouricemic tablets
- Placebo (Placebo Comparator): Generic name: Placebo Dosage form: Capsule Frequency: Two pills daily for 6 months
  Interventions: Combination Product: Placebo

INTERVENTIONS:
Combination Product: High-dose multi-vitamins with minerals — The high-dose multi-vitamins with minerals contained vitaminB1 0.72mg,vitamin B20.72mg,vitamin B12 1.35μg,folic acid 0.37mg,vitamin C 0.27mg,vitamin D 5.04μg,selenium 30.5μg per pill, respectively.
  Arms: High-dose multi-vitamins with minerals
Combination Product: Low-dose multi-vitamins with minerals — The low-dose multi-vitamins with minerals contained vitaminB1 0.72mg,vitamin B20.72mg,vitamin B12 1.35μg,folic acid 0.20mg,vitamin C 0.50mg,vitamin D 5.04μg,selenium 30.5μg per pill, respectively.
  Arms: Low-dose multi-vitamins with minerals
Combination Product: Hypouricemic tablets — The hypouricemic tablets contained skipjack,salvia and rosemary extract.
  Arms: Hypouricemic tablets
Combination Product: Placebo — The placebo tablets contained maltodextrin and tartrazine.
  Arms: Placebo

SUMMARY:
To evaluate the validity of multi-vitamin-and-minerals intervention on uric acid metabolism in hyperuricemic adults.

DETAILED DESCRIPTION:
Hyperuricemia is a type of metabolic diseases which caused by purine metabolic disorder and (or) uric acid excretion disorder. Uric acid is produced by cell metabolism and food purine metabolism as the end-point product. Excess alcohol and purine-rich food intake together with abnormal function of purine metabolic key enzyme are the main causes leading increasing serum level of uric acid. It has been a focus in nutritional area that a safer approach of preventing hyperuricemia by adjustment of nutritional intake. Primary studies found that proper supplement of microelements showed significant regulations in inflammation and oxidative stress induced by elevating level of uric acid. Therefore, this study will be conducted to test whether the supplement of multi-vitamins with minerals will lower the level of blood uric acid and improve the imbalance of microelement metabolism or not. The investigators will recruit 200 subjects of study who would be divided into four groups and accept intervention of high-dose multi-vitamins with minerals, low-dose multi-vitamins with minerals, hypouricemic tablets and placebo, respectively. After intervention of 3 or 6 months, serum uric acid and purine metabolism function will be detected. This study could provide references for illuminating the mechanism in purine metabolism and nutritional measures to control the pathological development of hyperuricemia.

ELIGIBILITY:
Inclusion Criteria:

* Under the dietary pattern of normal intake of purine, the level of serum uric acid is higher than 420μmol/L for male or 360μmol/L for female (not be detected twice at the same day).

Exclusion Criteria:

* Gouty arthritis, tophus or gouty nephropathy.
* Complications including diabetes, cardiovascular diseases (angina, myocardial infarction) and so on.
* Taken hypouricemic medicine in the last week before intervention, including allopurinol, benzbromarone, probenecid and so on.
* Had an operation in the past year.
* Malnutrition or severe obesity, BMI<18.5kg/m2 or >30.0 kg/m2.
* Mental diseases, tumor, hepatic cirrhosis or other diseases that may interfere with the intervention.
* Alcohol abuse (>80g/d)

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2018-01 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Serum uric acid | 1 year
  Level of uric acid was described in μmol/L

SECONDARY OUTCOMES:
Serum IL-1 | 1.5 years
  Inflammation condition，serum IL-1 was described in ng/l.
Serum IL-6 | 1.5 years
  Inflammation condition, level of IL-6 was described in ng/l
Serum IL-10 | 1.5 years
  Inflammation condition, level of IL-10 was described in ng/l
Serum TNF-α | 1.5 years
  Inflammation condition, level of TNF-α was described in ng/l
Serum CRP | 1.5 years
  Inflammation condition, level of CRP was described in mg/l
Serum c-peptide | 1.5 years
  Pancreas islets function, c-peptide was described in nmol/L.
Serum xanthine oxidase(XOD) activity | 1.5 years
  Purine metabolism function, XOD activity was described in in U/ml.
Serum phosphoribosyl pyrophosphate(PRPP) | 1.5 years
  Purine metabolism function, PRPP level was described in μmol/g Hb.
Serum Glutamine(Glu) | 1.5 years
  Purine metabolism function, Glu level was described in μmol/L.

CONTACTS AND LOCATIONS:
Overall Officials: Min Xia, Ph.D, Principal Investigator — Department of Nutrition,School of Public Health,Sun Yat-sen University
Locations (1):
- Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Do not share participants data